CLINICAL TRIAL: NCT03844165
Title: Fighting the Fatty Liver Pandemic: Developing Effective Protocols & Local Expertise to Deliver & Evaluate Diet/Lifestyle Interventions for Better Liver & Metabolic Health in India
Brief Title: Fighting Fatty Liver in India
Acronym: FFL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Population Health and Research Institute, Trivandrum, Kerala, india (Unknown); Holistic Health and Research Institute, Trivandrum, Kerala, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 137 1811
Record Dates: First submitted 2019-02-11; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: This is two-arm dietary interventional study that will be conducted through the Population Health and Research Institute, Trivandrum, India. Participants will be randomised to one of two study arms: diet change with yoga or yoga. We will aim to recruit 42 participants to each arm.
Who Masked: Investigator
Masking Description: The participant and study team will not be blinded to this allocation, although the scientist and radiology team will be blinded when analysing samples/scans.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet change (red rice) with yoga (Experimental): Following randomisation, participants are given a schedule of group and personal meetings and details of each session. Food for the diet (red rice and lentils) will be provided for those randomised to the diet arm. The study will last 16 weeks following start of the diet/yoga programme. There will be further visits to measure outcomes at week 8 and week 16. All participants in both arms will complete the same programme of Yoga sessions, organized and delivered by experienced practitioners under direction of Dr Leena Mohan at the Holistic Health and Research Institute.
  Interventions: Behavioral: Diet change (red rice); Behavioral: Yoga
- Yoga (Active Comparator): Following randomisation, participants are given a schedule of group and personal meetings and details of each session. The study will last 16 weeks following start of the diet/yoga programme. There will be further visits to measure outcomes at week 8 and week 16. All participants in both arms will complete the same programme of Yoga sessions, organized and delivered by experienced practitioners under direction of Dr Leena Mohan at the Holistic Health and Research Institute.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Diet change (red rice) — This interventions specifically aims to reduce liver inflammation, by replacing white rice in the diet with equal amounts of red rice and lentils. This will also enable for the research team to tests specific scientific hypotheses regarding the effects of diet on insulin resistance, liver pathology and the gut microbiome in NAFLD.
  Arms: Diet change (red rice) with yoga
Behavioral: Yoga — All 84 study participants take part in the yoga intervention. This is an intensive programme organized and delivered by experienced practitioners under direction of Dr Leena Mohan at the Holistic Health and Research Institute. This will evaluate whether physical activity alone improves metabolic health of the liver.

SUMMARY:
This study aims to build capacity in India by:

1. Developing tailored protocol methodologies for research including technical capability in imaging (MRI/S protocols & customised software), dietary intervention delivery, dietary evaluation, and biochemical analyses, using available local resources in Kerala.
2. Training and enhancing imaging skills of clinical radiographers in Kerala for research studies
3. Training local professionals and researchers in skills necessary to design, deploy and evaluate diet/lifestyle interventions, including patient engagement, in Kerala.

This study will deliver and evaluate a simple dietary intervention pilot study in the Kerala region in conjunction with local nutritionists, healthcare professionals and partner researchers at PHRI (Population Health and Research Institute, Trivandrum, Kerala, India).

DETAILED DESCRIPTION:
STUDY BACKGROUND INFORMATION AND RATIONALE

Non-alcoholic fatty liver disease (NAFLD):

With an estimated global prevalence of 25% among adults, NAFLD is now the commonest chronic liver disease; its progressive form, non-alcoholic steatohepatitis (NASH), has been estimated to affect 1.5%-6.5% of the population with associated increased risk of cirrhosis, hepatocellular carcinoma and liver-specific mortality. Considering the key association of fat accumulation within the liver, in particular diacyl glycerols, to the generation of whole body insulin resistance and development of type 2 diabetes, NAFLD has been considered a pre-diabetic state. NAFLD has been associated with excess risk of non-fatal and fatal cardiovascular events independently of established co-morbidities including type 2 diabetes, dyslipidemia and obesity. Individuals of South Asian ethnicity have significantly higher rates of NAFLD, abdominal obesity and cardiovascular disease than whites and ethnicity is a risk factor for NAFLD independent of diabetes, BMI, hypertension and hypercholesterolemia.

NAFLD problem in India:

Consistent with the global trend, the health and economic burdens of metabolic syndrome and NAFLD have risen in India. In 2011, India had 63 million individuals with type 2 diabetes and by 2030, that number is predicted to be a staggering 90 million. Insulin resistance (IR) has also been shown to be more prevalent in Indians compared with other ethnic groups and this has been correlated with NAFLD regardless of adiposity. Despite these links, there are a number of key differences between Indian NAFLD patients and those in the West: mean BMI is significantly lower in Indians and there is also a lower prevalence of hypertension, diabetes and metabolic syndrome in non-cirrhotic NAFLD patients.

Dietary influences on NAFLD:

Diet may be one of the key environmental factors that accounts for ethnic variation in susceptibility to NAFLD. However, there is currently a lack of research into specific dietary factors influencing susceptibility to NAFLD, in particular, with regards to macronutrients, and there are few evidence-based dietary interventions, beyond energy restriction to induce weight loss. Considering the effectiveness of a modest increase in protein content and a reduction in the glycaemic index (GI) in maintaining weight loss, we investigated the effects of a low GI diet on the liver and demonstrated that it did not increase liver fat content whereas an increase was seen with an isoenergetic high GI diet controlled for macronutrient content.

Diet has been found to influence the gut microbiome variably across human societies. Fibre encompassing a range of characteristics, is one of the fundamental components linking diet, the gut microbiome and fatty acid metabolism. The benefits of dietary fibre include improved glucose homeostasis and insulin sensitivity. Dietary fibres are at least partly fermented in the caecum and large intestine by the colonic microbiota resulting in some cases an increased production of short chain fatty acids (SCFAs) which regulate the balance between fatty acid synthesis, fatty acid oxidation and lipolysis in the body. The net result is a reduction in free fatty acid concentrations in plasma and a decrease in body weight. Dietary fibre overall is associated with greater gut microbiome diversity and we have recently shown that it is also associated with lower long-term weight gain.

ELIGIBILITY:
Inclusion criteria

* aged 18 years or over
* Male
* Able to give informed consent
* NAFLD diagnosis showing Fatty/echo-bright liver on ultrasound within past 3 months
* Able to attend yoga sessions
* Able to undergo MRI
* Consumer of at least 300g (uncooked weight) white rice per day (on average)
* No allergy to red rice or lentils
* Medically suitable for repeated blood sampling

Exclusion criteria

* Known or suspected cirrhosis on clinical/histological/radiological grounds
* Current or recent history of significant alcohol consumption (>14units per week)
* Other documented causes of chronic liver disease including:

  * Hepatitis B or C infection
  * Drug-induced liver disease
  * Alcohol-related liver disease
  * Autoimmune hepatitis
  * Wilson's disease, Haemachromatosis
  * Primary biliary cirrhosis, Primary Sclerosing Cholangitis
* Currently taking medication that can induce steatosis (corticosteroids, Amiodarone, Tamoxifen, Methotrexate)
* Evidence of any other unstable or untreated clinically significant immunological, endocrine, haematological, gastrointestinal, neurological, neoplastic or psychiatric disease
* *Female

  * A number of gender specific confounders (menstrual cycle, age etc) mean that mechanistic studies in small sample sizes are limited to men. The local cohort being used comprises males only.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — A number of gender specific confounders (menstrual cycle, age etc) mean that mechanistic studies in small sample sizes are limited to men. The local cohort being used comprises males only.
Enrollment: 84 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in liver fat | 1 year
  Measured by MRI, comparing liver fat pre- and post-intervention.

SECONDARY OUTCOMES:
Change in body composition | 1 year
  Measured by body fat % via bioimpedance
Change in body composition | 1 year
  Measured by BMI (kg/m2)
Change in insulin sensitivity | 1 year
  Measured by oral glucose tolerance test (OGTT)

CONTACTS AND LOCATIONS:
Locations (1):
- Population Health and Research Institute, Trivandrum, Kerala, India

IPD SHARING:
Plan to Share IPD: Undecided